CLINICAL TRIAL: NCT04567134
Title: Clostridioides Difficile Infection - a Prospective Nationwide Epidemiologic Study in Korea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Korean Center for Disease Control and Prevention (Other Government); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: HYUH 2020-06-046
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Clostridium Difficile Infection
Keywords: clostridium difficile; incidence
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — C. difficile isolates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our objective of this study is to derive a real incidence of CDI in tertiary hospitals located through Korean peninsula. In order to get a close value to the truth, the study is planned to co-perform with a national study which was proposed in evaluation process to include more hospitals. Along with the incidence of CDI, clinical characteristics and outcome of CDI will be examined and microbiologic characteristics of C. difficile isolates from CDI patients are studied.

ELIGIBILITY:
Inclusion Criteria:

* aged older than 19 years
* more than 3 times of unformed stools passage per day
* positive results of toxin gene test: GDH (+) + PCR (+), GDH (+) + toxin (+), or PCR (+) + toxin (+)
* agree with informed consent

Exclusion Criteria:

* less than 3 times of unformed stool passage per day
* use of oral metronidazole or vancomycin more than 24 hours before enrollment
* use of laxative before enrollment
* recurrent episode of CDI
* disagree with study protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who admitted at the tertiary hospitals in Korea and and diagnosed as Clostridioides difficile infection will be selected.
  The tertiary hospitals located in Seoul-si, Gyeonggi-do, Pusan-si, Daegu-si, Jeollanam-do, Jeollabuk-do, and Chungcheongbuk-do. These hospitals distributes all over the country.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of CDI | through Oct 2020 to Dec 2021
  Incidence of CDI among hospitalized adults per 100,000 patient*days/10,000 patient*admission in enrolled tertiary hospitals.

SECONDARY OUTCOMES:
mortality rate | through Oct 2020 to May 2022
  Proportion of CDI cases who died during the 60-day follow-up period
recurrence rate | through Oct 2020 to May 2022
  Proportion of CDI cases with recurrence/reinfection between Day 14 and Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Hyunjoo Pai, M.D., Ph.D., Study Chair — Hanyang University College of Medicine